CLINICAL TRIAL: NCT00524901
Title: An Open Label Study to Evaluate the Effect of Intravenous Erythropoietin on Erythropoietin Receptor Signaling and Markers for Apoptosis, Myocardial Damage and Renal Dysfunction in Patients Undergoing Coronary Artery Bypass Graft (CABG) Surgery
Brief Title: Study of the Use of a Single Dose of Erythropoietin to Treat Acute Myocardial Ischemia
Acronym: DREAM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Willem-Peter Theodoor Ruifrok, MD, PhD, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WTR-ECG-2
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: CABG; Coronary Artery Disease
Keywords: Apoptosis; CABG; Coronary Artery Disease; Three Vessel Disease; Erythropoietin; EPO-receptor signaling
MeSH Terms: conditions — Coronary Artery Disease | interventions — Epoetin Alfa; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 25 patients undergoing CABG for three vessel disease, receiving a single dose of erythropoietin periprocedural.
  Interventions: Drug: Epoetin alpha
- 2 (Placebo Comparator): 25 patients undergoing CABG for three vessel disease, receiving placebo (NaCl 0.9%) periprocedural.
  Interventions: Drug: NaCl 0.9%

INTERVENTIONS:
Drug: Epoetin alpha — A single dose of epoetin alpha during CABG for three vessel disease, 60.000 IU intravenously.
  Other Names: Eprex
  Arms: 1
Drug: NaCl 0.9% — A single dose of NaCl 0.9% during CABG for three vessel disease, 1 ml intravenously.
  Other Names: Saline
  Arms: 2

SUMMARY:
This is a phase 2 study that evaluates the effect of intravenous administration of a bolus EPO on the activation of EPOR-signal transduction cascades and myocardial apoptosis during cardiopulmonary bypass surgery. Human atrial and ventricular tissue will be collected during CABG surgery for 3-vessel disease for the assay of EPOR signaling and apoptosis. Two atrial specimens will be collected before and at the end of cardiopulmonary bypass (CPB). Concomitantly, two transmural ventricular biopsies will be obtained, at the start and at the end of CPB. Immediately after obtaining the first atrial biopsy, one bolus of EPO will be administered intravenously. The atrial tissue will be split and appropriate sections will be frozen for determination of baseline expression or activity of a number of molecules including Erk1/2, STAT5, Akt and caspase-3 or embedded in paraffin for immunohistochemistry. Ventricular tissue will only be processed for immunohistochemistry. Additionally, plasma will be collected before the procedure and for up to 30 days post-procedure to examine release of markers of both myocardial ischemia and stress (CK-MB, Troponin T and NT-proBNP) and renal dysfunction (cystatin C, creatinine for eGFR). Before initializing the randomised study, a pilot study will be performed with 5 subjects that will not be treated to evaluate the feasibility of myocardial sample collection. Initiation of the randomised study will only commence if baseline activity of EPOR-STC can be determined in the atrial tissue and caspase-3 positive cells can be identified in the second ventricular biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Before any study-specific procedure, including assessments for screening, the appropriate written informed consent must be obtained.
* Man or woman 18 to 80 years of age .
* Undergoing a planned, elective cardiopulmonary bypass operation for the first time for 3-vessel coronary artery disease with an anticipated aortic cross clamp time of approximately 40 minutes and a total bypass time of approximately 90 minutes.
* Hemoglobin (Hb) concentration ≥7.4 mmol/l and ≤9.9 mmol/l within 7 days prior to CABG surgery and no major acute blood loss since this Hb determination.

Exclusion Criteria:

* An unstable medical condition, defined as having been hospitalized for a non-cardiac condition within 4 weeks of screening, major surgery within 24 weeks of screening, or otherwise unstable in the judgment of the investigator (e.g., at risk of complications or adverse events unrelated to study participation).
* Left ventricular ejection fraction (LVEF) < 40%.
* Clinical history of chronic kidney disease (CKD) (at any point prior to registration) defined as serum creatinine >105 μmol/l for all females, >130 μmol/l for black males, and >115 μmol/l for non-black males.
* Atrial fibrillation, paroxysmal atrial fibrillation or atrial flutter.
* Clinically significant abnormality in chemistry, hematology, or urinalysis parameters performed within the screening period.
* Current symptoms of polyurea, polydipsia, or increased thirst.
* Grand mal seizure within 1 year of enrollment.
* Poorly controlled hypertension, defined as systolic blood pressure (SBP) > 180 mmHg or diastolic blood pressure (DBP) > 105 mmHg on day of CABG surgery.
* Use of any erythropoietic protein (e.g., rHuEPO; Procrit®, Eprex®, Neorecormon®, Epogen®, Aranesp®) within 12 weeks of enrolment.
* Positive pregnancy test or known to be pregnant at the time of screening.
* Recent (within 3 months) history of alcohol or illicit drug abuse disorder, based on self-report.
* Severe uncorrected valvular disease (including pulmonary and tricuspid) or left ventricular outflow obstruction which, in the opinion of the investigator, requires surgery.
* Pulmonary hypertension, defined as a pulmonary artery pressure > 30 mmHg at rest.
* Participation in any investigational device or drug trial(s) or receiving other investigational agent(s) within 30 days.
* Known positive for HIV antibodies, hepatitis B surface antigen, or hepatitis C antibodies.
* Any condition (e.g., unsuitable anatomy of the atrium; psychiatric illness; etc.) or situation that, in the investigator's opinion, could put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-09; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The increase from baseline between EPO and saline treated subjects in activity of EPOR-STC including but not limited to, phospho Erk1/2, phospho Akt, activated caspase-3, and activated STAT5 in the second atrial biopsy. | 2 hours

SECONDARY OUTCOMES:
Difference in apoptosis between atrial and ventricular specimens at the end of CPB, defined as the number of TUNEL and activated caspase-3 positive cells per high power field. | 2 hours
Difference between EPO- and saline treated subjects in TUNEL and active caspase-3 positive cells in ventricular and atrial biopsies. | 2 hours
Difference in AUC for CK-MB, Troponin T, NT-proBNP, and cystatin C between EPO- and saline treated patients. | 30 days
Subject incidence rates of adverse events. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: W. H. van Gilst, Prof, dr, Study Chair — University Medical Center Groningen, Dept. of Exprimental Cardiology; W. T. Ruifrok, MD, Principal Investigator — University Medical Center Groningen, Dept. of Experimental Cardiology; B. D. Westenbrink, MD, Principal Investigator — University Medical Center Groningen, Dept. of Experimental Cardiology; A. H. Epema, dr, MD, Principal Investigator — University Medical Center Groningen, Dept. of Anaesthesiology; H. E. Mungroop, dr, MD, Principal Investigator — University Medical Center Groningen, Dept. of Anaesthesiology; P. W. Boonstra, Prof, dr, MD, Principal Investigator — University Medical Center Groningen, Dept. of Cardiothoracic Surgery; R. A. de Boer, dr, MD, Principal Investigator — University Medical Center Groningen, Dept of Cardiology; D. J. van Veldhuisen, Prof, dr, MD, Study Director — University Medical Center Groningen, Dept. of Cardiology
Locations (1):
- University Medical Center Groningen, Dept. of Cardiology, Groningen, Provincie Groningen, Netherlands